CLINICAL TRIAL: NCT01728402
Title: Pathogenesis of Acute Leukemia, Lymphoproliferative Disorders, and Myeloproliferative Disorders
Brief Title: Pathogenesis of Hematologic Malignancies
Status: Enrolling by invitation | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marc Loriaux, Associate Professor, OHSU Knight Cancer Institute
Other Study IDs: IRB00004422; 5R21CA159265 (NIH)
Record Dates: First submitted 2012-11-13; First posted 2012-11-19 (Estimated); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Acute Leukemia; Lymphoproliferative Disorders; Myeloproliferative Disorders; Myelodysplastic Syndromes
MeSH Terms: conditions — Lymphoproliferative Disorders; Myeloproliferative Disorders; Myelodysplastic Syndromes | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood Draw
  Interventions: Procedure: blood draw, bone marrow procedure, or tissue biopsy

INTERVENTIONS:
Procedure: blood draw, bone marrow procedure, or tissue biopsy

SUMMARY:
The cause of blood and bone marrow cancers is poorly understood; however, most research focuses on how cancer cells grow and develop. Because the causes of these cancers are unknown, current treatments may be unnecessarily harsh and often do not provide a cure. Identifying the causes of blood cancers would allow for the development of treatments that are more likely to provide a cure. To find the causes of blood and bone marrow cancers, we will look for specific cancer cell abnormalities that are responsible for cancer cell growth. We will then look to see if drugs that can reverse these abnormalities can kill cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed diagnosis of AL, LPD, MDS, or MPD
* Male or female of all ages
* Willing and able to sign informed consent
* Willing guardian consent for participants under 18 years of age

Exclusion Criteria:

* No suspected or confirmed diagnosis of acute leukemias (AL), lymphoproliferative disorders (LPD), myelodysplastic syndromes (MDS), or myeloproliferative diseases (MPD)

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of any age with a diagnosis or suspected diagnosis of a blood or bone marrow cancer may be a part of this study. The provider who will perform the blood draw, bone marrow aspirate, or biopsy as part of the patient's routine care will identify possible participants from their clinic schedule or patient list, give them information about what would be involved in participating in the study including possible risks, and ask if they are interested in participating.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2008-09

PRIMARY OUTCOMES:
Identify and determine the frequency of mutations causing aberrant signaling pathway function in patients with acute leukemias (AL), lymphoproliferative disorders (LPD), myelodysplastic syndromes (MDS), and myeloproliferative neoplasms (MPN) | After laboratory analyses are complete. Lab samples are collected at the time of a scheduled blood draw, bone marrow procedure, tissue biopsy, or other visit for usual medical care
  Integrated functional genomics studies (whole genome sequencing, RNAi, proteomics, drug sensitivity, expression profiling) will be used to identify aberrant signaling pathways that contribute to the formation of hematologic malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Loriaux, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States